CLINICAL TRIAL: NCT05008211
Title: Effectiveness of an Information-Motivation-Behavioral Skills Model-based Intervention on Adherence to Domiciliary Non-invasive Ventilation of Patients With Chronic Hypercapnic Respiratory Failure: A Randomized Controlled Study
Brief Title: Information-Motivation-Behavioral Skills Model-based Intervention to Domiciliary Non-invasive Ventilation of Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: University Grants Committee, Hong Kong (Other Government); Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Prof. Yu, Doris Sau Fung, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IMB-NIV-CHRF
Record Dates: First submitted 2021-08-09; First posted 2021-08-17 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Hypercapnic Respiratory Failure; Noninvasive Ventilation
Keywords: Chronic Hypercapnic Respiratory Failure; Chronic Obstructive Pulmonary Disease; Noninvasive Ventilation; hospital admission; respiratory insufficiency
MeSH Terms: conditions — Respiratory Insufficiency; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): There will be a respiratory team, same as the usual care, responsible for patients requiring domiciliary NIV in the intervention group.
  The IMB model-based intervention of this study is a six-week program consisted of a one-hour face-to-face home visit in the first week, two 20-minute telephone follow-ups in the second and fourth weeks, and a half-hour face-to-face follow-up at hospital in the sixth week, and a telephone consultation hotline during office hours.
  There are three major components including information, motivation and behavioral skill interventions as proposed by the IMB model and will be deliberately arranged in the different sessions.
  Interventions: Other: Information-Motivation-Behavioral skills (IMB) model-based intervention
- Control - usual care (Placebo Comparator): There is a respiratory team of health care professionals responsible for patients requiring domiciliary NIV. The team is led by a Medical Consultant and with respiratory nurse(s) as team members who are responsible for assisting patients or their family to initiate domiciliary NIV and teaching the relevant technical skills. The nurse will provide an one-hour face-to-face session to introduce the choices of domiciliary NIV and teach the patient or his/her family on how to operate and maintain the ventilator, interface and accessories, and also how to handle the common problems such as leakage and pressure sore in hospital before discharge. Commercial leaflet or booklet according to the choice of ventilator with information of the ventilator, interface, accessories and the ventilator company will be provided to the patient.
  Interventions: Other: Control - usual care

INTERVENTIONS:
Other: Information-Motivation-Behavioral skills (IMB) model-based intervention — A six-week programme
  Arms: Intervention
Other: Control - usual care — he nurse will provide an one-hour face-to-face session to introduce the choices of domiciliary NIV and teach the patient or his/her family on how to operate and maintain the ventilator, interface and accessories, and also how to handle the common problems
  Arms: Control - usual care

SUMMARY:
Domiciliary non-invasive ventilation (NIV) is a standard care for improving survival rates of selected patients with chronic hypercapnic respiratory failure (CHRF) and to improve the patients' hypercapnia, sleep quality, health-related quality of life (QoL). Adherence is an important factor affecting clinical effectiveness of domiciliary NIV. Our previous study has noted the associations between poor domiciliary NIV adherence and increased number of clinical adverse events (p = 0.004) and increased hospitalization requiring acute NIV salvage (p = 0.042). However, there are very limited studies on adherence to domiciliary NIV in patients with CHRF. The only interventional study was a single-group pre-test post-test study and lack of a theoretical framework for guiding the intervention. This study is employing an Information-Motivation-Behavioral skills (IMB) model-based intervention to improve inhalation adherence in a group of chronic obstructive pulmonary disease (COPD) patients.

DETAILED DESCRIPTION:
The study design is a multi-center, 2-arm single-blind randomized controlled trial. The intervention group will receive an Information-Motivation-Behavioral (IMB) model-based intervention while the control group will receive the usual care.

Usual Care: There is a respiratory team of health care professionals responsible for patients requiring domiciliary non-invasive ventilation (NIV). The team is led by a Medical Consultant and with respiratory nurse(s) as team members who are responsible for assisting patients or their family to initiate domiciliary NIV and teaching the relevant technical skills. The nurse will provide an one-hour face-to-face session to introduce the choices of domiciliary NIV and teach the patient or his/her family on how to operate and maintain the ventilator, interface and accessories, and also how to handle the common problems such as leakage and pressure sore in hospital before discharge. Commercial leaflet or booklet according to the choice of ventilator with information of the ventilator, interface, accessories and the ventilator company will be provided to the patient.

Intervention:

There will be a respiratory team, same as the usual care, responsible for patients requiring domiciliary NIV in the intervention group. The IMB model-based intervention of this study is a six-week program consisted of a one-hour face-to-face home visit in the first week, two 20-minute telephone follow-ups in the second and fourth weeks, and a half-hour face-to-face follow-up at hospital in the sixth week, and a telephone consultation hotline during office hours.

ELIGIBILITY:
Inclusion Criteria:

* (1) CHRF (i.e., PaCO2 ≥ 7 kPa or 52.5 mmHg) for at least 4 weeks, and
* (2) using domiciliary NIV for ≥ 4 weeks, and
* (3) non-adherer (i.e., used domiciliary NIV for < 4 hours per night or < 70% of days or with a mean daily use < 5 hours per day in the last 2 weeks)

Exclusion Criteria:

* (1) known psychiatric disorders except anxiety and depression; or
* (2) diseases limiting life expectancy to ≤ one year; or
* (3) active malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Domiciliary NIV adherence | baseline
  the records from the software fitted on the subject's NIV machine for the past two weeks will be reviewed to determine adherence or non-adherence, and assessed for the percentage of days with usage of at least 4 hours per night and the mean of daily use.
Domiciliary NIV adherence | 3rd month
  the records from the software fitted on the subject's NIV machine for the past two weeks will be reviewed to determine adherence or non-adherence, and assessed for the percentage of days with usage of at least 4 hours per night and the mean of daily use.
Domiciliary NIV adherence | 6th month
  the records from the software fitted on the subject's NIV machine for the past two weeks will be reviewed to determine adherence or non-adherence, and assessed for the percentage of days with usage of at least 4 hours per night and the mean of daily use.
Domiciliary NIV adherence | 12th month
  the records from the software fitted on the subject's NIV machine for the past two weeks will be reviewed to determine adherence or non-adherence, and assessed for the percentage of days with usage of at least 4 hours per night and the mean of daily use.

SECONDARY OUTCOMES:
Venous bicarbonate (HCO3-) level | baseline
  estimation for level of hypercapnia
Venous bicarbonate (HCO3-) level | 3rd month
  estimation for level of hypercapnia
Venous bicarbonate (HCO3-) level | 6th month
  estimation for level of hypercapnia
Chinese Pittsburgh Sleep Quality Index (CPSQI) | baseline
  19-item self-reported measures assess the participant's sleep quality over last month. Seven component scores including subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, sleep medication, and daytime dysfunction can be obtained from the items. The component scores range from 0 (no problem) to 3 (severe problem) and the overall score ranges from 0 to 21 with a higher score indicating a poorer sleep quality.
Chinese Pittsburgh Sleep Quality Index (CPSQI) | 3rd month
  19-item self-reported measures assess the participant's sleep quality over last month. Seven component scores including subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, sleep medication, and daytime dysfunction can be obtained from the items. The component scores range from 0 (no problem) to 3 (severe problem) and the overall score ranges from 0 to 21 with a higher score indicating a poorer sleep quality.
Chinese Pittsburgh Sleep Quality Index (CPSQI) | 6th month
  19-item self-reported measures assess the participant's sleep quality over last month. Seven component scores including subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, sleep medication, and daytime dysfunction can be obtained from the items. The component scores range from 0 (no problem) to 3 (severe problem) and the overall score ranges from 0 to 21 with a higher score indicating a poorer sleep quality.
Chinese Pittsburgh Sleep Quality Index (CPSQI) | 12th month
  19-item self-reported measures assess the participant's sleep quality over last month. Seven component scores including subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, sleep medication, and daytime dysfunction can be obtained from the items. The component scores range from 0 (no problem) to 3 (severe problem) and the overall score ranges from 0 to 21 with a higher score indicating a poorer sleep quality.
Chinese Severe Respiratory Insufficiency questionnaire (CSRI) | baseline
  49 items assess the participants's health-related quality of life (QoL) from completely untrue, mostly untrue, sometimes true , mostly true, always true. The scores will be transformed between 0 and 100 with higher values indicating a better health-related quality of life.
Chinese Severe Respiratory Insufficiency questionnaire (CSRI) | 3rd month
  49 items assess the participants's health-related quality of life (QoL) from completely untrue, mostly untrue, sometimes true , mostly true, always true. The scores will be transformed between 0 and 100 with higher values indicating a better health-related quality of life.
Chinese Severe Respiratory Insufficiency questionnaire (CSRI) | 6th month
  49 items assess the participants's health-related quality of life (QoL) from completely untrue, mostly untrue, sometimes true , mostly true, always true. The scores will be transformed between 0 and 100 with higher values indicating a better health-related quality of life.
Chinese Severe Respiratory Insufficiency questionnaire (CSRI) | 12th month
  49 items assess the participants's health-related quality of life (QoL) from completely untrue, mostly untrue, sometimes true , mostly true, always true. The scores will be transformed between 0 and 100 with higher values indicating a better health-related quality of life.
Hospital admissions and survival rate | baseline
  record the number of hospital admissions
Hospital admissions and survival rate | 12th month
  record the number of hospital admissions

CONTACTS AND LOCATIONS:
Overall Officials: Doris SF Yu, PhD, Principal Investigator — School of Nursing, LKS Faculty of Medicine, HKU; Henry Poon, PhD, Study Chair — United Christian Hospital
Locations (1):
- Department of Medicine and Geriatrics, United Christian Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Only study investigators and research assistants involved in the study will have access to the data.

REFERENCES:
- [Result] Hormann C, Baum M, Putensen C, Mutz NJ, Benzer H. Biphasic positive airway pressure (BIPAP)--a new mode of ventilatory support. Eur J Anaesthesiol. 1994 Jan;11(1):37-42. PMID 8143712
- [Result] Chu CM, Yu WC, Tam CM, Lam CW, Hui DS, Lai CK; Hong Kong Home Ventilation Registry; Hong Kong Thoracic Society. Home mechanical ventilation in Hong Kong. Eur Respir J. 2004 Jan;23(1):136-41. doi: 10.1183/09031936.03.00017803. PMID 14738245
- [Result] Simonds AK. Home Mechanical Ventilation: An Overview. Ann Am Thorac Soc. 2016 Nov;13(11):2035-2044. doi: 10.1513/AnnalsATS.201606-454FR. PMID 27560387
- [Result] Cheng SL, Chan VL, Chu CM. Compliance with home non-invasive ventilation. Respirology. 2012 May;17(4):735-6. doi: 10.1111/j.1440-1843.2012.02169.x. PMID 22420583
- [Result] Motor Neurone Disease: The Use of Non-Invasive Ventilation in the Management of Motor Neurone Disease [Internet]. London: National Institute for Health and Clinical Excellence (NICE); 2010 Jul. Available from http://www.ncbi.nlm.nih.gov/books/NBK65383/ PMID 22171400
- [Result] Simonds AK, Elliott MW. Outcome of domiciliary nasal intermittent positive pressure ventilation in restrictive and obstructive disorders. Thorax. 1995 Jun;50(6):604-9. doi: 10.1136/thx.50.6.604. PMID 7638799
- [Result] Leger P, Bedicam JM, Cornette A, Reybet-Degat O, Langevin B, Polu JM, Jeannin L, Robert D. Nasal intermittent positive pressure ventilation. Long-term follow-up in patients with severe chronic respiratory insufficiency. Chest. 1994 Jan;105(1):100-5. doi: 10.1378/chest.105.1.100. PMID 8275718
- [Result] Mehta S, Hill NS. Noninvasive ventilation. Am J Respir Crit Care Med. 2001 Feb;163(2):540-77. doi: 10.1164/ajrccm.163.2.9906116. No abstract available. PMID 11179136
- [Result] Shneerson JM, Simonds AK. Noninvasive ventilation for chest wall and neuromuscular disorders. Eur Respir J. 2002 Aug;20(2):480-7. doi: 10.1183/09031936.02.00404002. PMID 12212984
- [Result] Meecham Jones DJ, Paul EA, Jones PW, Wedzicha JA. Nasal pressure support ventilation plus oxygen compared with oxygen therapy alone in hypercapnic COPD. Am J Respir Crit Care Med. 1995 Aug;152(2):538-44. doi: 10.1164/ajrccm.152.2.7633704.
- [Result] Elliott MW, Mulvey DA, Moxham J, Green M, Branthwaite MA. Domiciliary nocturnal nasal intermittent positive pressure ventilation in COPD: mechanisms underlying changes in arterial blood gas tensions. Eur Respir J. 1991 Oct;4(9):1044-52. PMID 1756837
- [Result] Ambrosino N, Montagna T, Nava S, Negri A, Brega S, Fracchia C, Zocchi L, Rampulla C. Short term effect of intermittent negative pressure ventilation in COPD patients with respiratory failure. Eur Respir J. 1990 May;3(5):502-8. PMID 2376246
- [Result] Duiverman ML, Wempe JB, Bladder G, Vonk JM, Zijlstra JG, Kerstjens HA, Wijkstra PJ. Two-year home-based nocturnal noninvasive ventilation added to rehabilitation in chronic obstructive pulmonary disease patients: a randomized controlled trial. Respir Res. 2011 Aug 23;12(1):112. doi: 10.1186/1465-9921-12-112. PMID 21861914
- [Result] Suraj KP, Jyothi E, Rakhi R. Role of Domiciliary Noninvasive Ventilation in Chronic Obstructive Pulmonary Disease Patients Requiring Repeated Admissions with Acute Type II Respiratory Failure: A Prospective Cohort Study. Indian J Crit Care Med. 2018 Jun;22(6):397-401. doi: 10.4103/ijccm.IJCCM_61_18. PMID 29962738
- [Result] Blankenburg T, Benthin C, Pohl S, Bramer A, Kalbitz F, Lautenschlager C, Schutte W. Survival of Hypercapnic Patients with COPD and Obesity Hypoventilation Syndrome Treated with High Intensity Non Invasive Ventilation in the Daily Routine Care. Open Respir Med J. 2017 Jun 30;11:31-40. doi: 10.2174/1874306401711010031. eCollection 2017. PMID 28839495
- [Result] Duiverman ML, Windisch W, Storre JH, Wijkstra PJ. The role of NIV in chronic hypercapnic COPD following an acute exacerbation: the importance of patient selection? Ther Adv Respir Dis. 2016 Apr;10(2):149-57. doi: 10.1177/1753465815624645. Epub 2016 Jan 8. PMID 26746384
- [Result] Kohnlein T, Windisch W, Kohler D, Drabik A, Geiseler J, Hartl S, Karg O, Laier-Groeneveld G, Nava S, Schonhofer B, Schucher B, Wegscheider K, Criee CP, Welte T. Non-invasive positive pressure ventilation for the treatment of severe stable chronic obstructive pulmonary disease: a prospective, multicentre, randomised, controlled clinical trial. Lancet Respir Med. 2014 Sep;2(9):698-705. doi: 10.1016/S2213-2600(14)70153-5. Epub 2014 Jul 24. PMID 25066329
- [Result] Dreher M, Storre JH, Schmoor C, Windisch W. High-intensity versus low-intensity non-invasive ventilation in patients with stable hypercapnic COPD: a randomised crossover trial. Thorax. 2010 Apr;65(4):303-8. doi: 10.1136/thx.2009.124263. PMID 20388753
- [Result] McEvoy RD, Pierce RJ, Hillman D, Esterman A, Ellis EE, Catcheside PG, O'Donoghue FJ, Barnes DJ, Grunstein RR; Australian trial of non-invasive Ventilation in Chronic Airflow Limitation (AVCAL) Study Group. Nocturnal non-invasive nasal ventilation in stable hypercapnic COPD: a randomised controlled trial. Thorax. 2009 Jul;64(7):561-6. doi: 10.1136/thx.2008.108274. Epub 2009 Feb 12. PMID 19213769
- [Result] Altintas N. Update: Non-Invasive Positive Pressure Ventilation in Chronic Respiratory Failure Due to COPD. COPD. 2016;13(1):110-21. doi: 10.3109/15412555.2015.1043520. Epub 2015 Sep 29. PMID 26418151
- [Result] Murphy PB, Rehal S, Arbane G, Bourke S, Calverley PMA, Crook AM, Dowson L, Duffy N, Gibson GJ, Hughes PD, Hurst JR, Lewis KE, Mukherjee R, Nickol A, Oscroft N, Patout M, Pepperell J, Smith I, Stradling JR, Wedzicha JA, Polkey MI, Elliott MW, Hart N. Effect of Home Noninvasive Ventilation With Oxygen Therapy vs Oxygen Therapy Alone on Hospital Readmission or Death After an Acute COPD Exacerbation: A Randomized Clinical Trial. JAMA. 2017 Jun 6;317(21):2177-2186. doi: 10.1001/jama.2017.4451. PMID 28528348
- [Result] Struik FM, Lacasse Y, Goldstein RS, Kerstjens HA, Wijkstra PJ. Nocturnal noninvasive positive pressure ventilation in stable COPD: a systematic review and individual patient data meta-analysis. Respir Med. 2014 Feb;108(2):329-37. doi: 10.1016/j.rmed.2013.10.007. Epub 2013 Oct 14. PMID 24157199
- [Result] Borel JC, Pepin JL, Pison C, Vesin A, Gonzalez-Bermejo J, Court-Fortune I, Timsit JF. Long-term adherence with non-invasive ventilation improves prognosis in obese COPD patients. Respirology. 2014 Aug;19(6):857-65. doi: 10.1111/resp.12327. Epub 2014 Jun 9. PMID 24912564
- [Result] Dretzke J, Moore D, Dave C, Mukherjee R, Price MJ, Bayliss S, Wu X, Jordan RE, Turner AM. The effect of domiciliary noninvasive ventilation on clinical outcomes in stable and recently hospitalized patients with COPD: a systematic review and meta-analysis. Int J Chron Obstruct Pulmon Dis. 2016 Sep 16;11:2269-2286. doi: 10.2147/COPD.S104238. eCollection 2016. PMID 27698560
- [Result] Farrero E, Prats E, Manresa F, Escarrabill J. Outcome of non-invasive domiciliary ventilation in elderly patients. Respir Med. 2007 Jun;101(6):1068-73. doi: 10.1016/j.rmed.2006.10.005. Epub 2006 Nov 28. PMID 17126543
- [Result] Callegari J, Magnet FS, Taubner S, Berger M, Schwarz SB, Windisch W, Storre JH. Interfaces and ventilator settings for long-term noninvasive ventilation in COPD patients. Int J Chron Obstruct Pulmon Dis. 2017 Jun 28;12:1883-1889. doi: 10.2147/COPD.S132170. eCollection 2017. PMID 28721033
- [Result] Chang AY, Marsh S, Smith N, Neill A. Long-term community non-invasive ventilation. Intern Med J. 2010 Nov;40(11):764-71. doi: 10.1111/j.1445-5994.2010.02171.x. PMID 20059598
- [Result] Ulger AF, Poyraz B, Gulec Balbay E, Binay S. Our experience of 200 patients: usage and maintenance of long-term oxygen therapy and non-invasive ventilation devices at home. Int J Clin Exp Med. 2014 Jan 15;7(1):170-6. eCollection 2014. PMID 24482704
- [Result] Gale NK, Jawad M, Dave C, Turner AM. Adapting to domiciliary non-invasive ventilation in chronic obstructive pulmonary disease: a qualitative interview study. Palliat Med. 2015 Mar;29(3):268-77. doi: 10.1177/0269216314558327. Epub 2014 Dec 18. PMID 25524958
- [Result] Ennis J, Rohde K, Chaput JP, Buchholz A, Katz SL. Facilitators and Barriers to Noninvasive Ventilation Adherence in Youth with Nocturnal Hypoventilation Secondary to Obesity or Neuromuscular Disease. J Clin Sleep Med. 2015 Dec 15;11(12):1409-16. doi: 10.5664/jcsm.5276. PMID 26235150
- [Result] Mansell SK, Cutts S, Hackney I, Wood MJ, Hawksworth K, Creer DD, Kilbride C, Mandal S. Using domiciliary non-invasive ventilator data downloads to inform clinical decision-making to optimise ventilation delivery and patient compliance. BMJ Open Respir Res. 2018 Mar 3;5(1):e000238. doi: 10.1136/bmjresp-2017-000238. eCollection 2018. PMID 29531743
- [Result] Mayberry LS, Osborn CY. Empirical validation of the information-motivation-behavioral skills model of diabetes medication adherence: a framework for intervention. Diabetes Care. 2014;37(5):1246-53. doi: 10.2337/dc13-1828. Epub 2014 Mar 5. PMID 24598245
- [Result] Cooperman NA, Richter KP, Bernstein SL, Steinberg ML, Williams JM. Determining Smoking Cessation Related Information, Motivation, and Behavioral Skills among Opiate Dependent Smokers in Methadone Treatment. Subst Use Misuse. 2015 Apr;50(5):566-81. doi: 10.3109/10826084.2014.991405. Epub 2015 Jan 5. PMID 25559697
- [Result] Nelson LA, Wallston KA, Kripalani S, LeStourgeon LM, Williamson SE, Mayberry LS. Assessing barriers to diabetes medication adherence using the Information-Motivation-Behavioral skills model. Diabetes Res Clin Pract. 2018 Aug;142:374-384. doi: 10.1016/j.diabres.2018.05.046. Epub 2018 Jun 4. PMID 29879495
- [Result] Malatesha G, Singh NK, Bharija A, Rehani B, Goel A. Comparison of arterial and venous pH, bicarbonate, PCO2 and PO2 in initial emergency department assessment. Emerg Med J. 2007 Aug;24(8):569-71. doi: 10.1136/emj.2007.046979. PMID 17652681
- [Result] Tsai PS, Wang SY, Wang MY, Su CT, Yang TT, Huang CJ, Fang SC. Psychometric evaluation of the Chinese version of the Pittsburgh Sleep Quality Index (CPSQI) in primary insomnia and control subjects. Qual Life Res. 2005 Oct;14(8):1943-52. doi: 10.1007/s11136-005-4346-x. PMID 16155782
- [Result] Ho RT, Fong TC. Factor structure of the Chinese version of the Pittsburgh sleep quality index in breast cancer patients. Sleep Med. 2014 May;15(5):565-9. doi: 10.1016/j.sleep.2013.10.019. Epub 2014 Feb 18. PMID 24759325
- [Result] Cheung LM, Wong WS. The effects of insomnia and internet addiction on depression in Hong Kong Chinese adolescents: an exploratory cross-sectional analysis. J Sleep Res. 2011 Jun;20(2):311-7. doi: 10.1111/j.1365-2869.2010.00883.x. Epub 2010 Aug 31. PMID 20819144
- [Result] Wong WS, Fielding R. Prevalence of insomnia among Chinese adults in Hong Kong: a population-based study. J Sleep Res. 2011 Mar;20(1 Pt 1):117-26. doi: 10.1111/j.1365-2869.2010.00822.x. PMID 20408932
- [Result] Chen R, Guan L, Wu W, Yang Z, Li X, Luo Q, Liang Z, Wang F, Guo B, Huo Y, Yang Y, Zhou L. The Chinese version of the Severe Respiratory Insufficiency questionnaire for patients with chronic hypercapnic chronic obstructive pulmonary disease receiving non-invasive positive pressure ventilation. BMJ Open. 2017 Aug 28;7(8):e017712. doi: 10.1136/bmjopen-2017-017712. PMID 28851800
- [Derived] Yu DSF, Li PW, Lau JC, Cheung PSA, Ip M, Cheng SLL, Poon HCL, Iris Lee FK. Health Communication and Adherence to Noninvasive Ventilation in Chronic Hypercapnic Respiratory Failure: A Randomized Clinical Trial. JAMA Netw Open. 2024 Dec 2;7(12):e2451614. doi: 10.1001/jamanetworkopen.2024.51614. PMID 39724376
- See also: Cheung PS, Chu CM. Non-invasive ventilation for COPD hospital and home use. The Hong Kong Medical Diary 2016; 21(9): 21-3. — http://www.fmshk.org/database/hkmd/hkmd201609.pdf
- See also: Comer DM. An update on domiciliary non-invasive ventilation. J Pulm Respir Med 2014; 5: 234. doi:10.4172/2161-105x.1000234 — https://www.hilarispublisher.com/open-access/an-update-on-domiciliary-noninvasive-ventilation-2161-105X.1000234.pdf
- See also: Sabate E. Adherence to long-term therapies: Evidence for action. Geneva, Switzerland: World Health Organization, 2003. — https://apps.who.int/iris/bitstream/handle/10665/42682/9241545992.pdf
- See also: Fisher WA, Fisher JD, Harman J. The Information-Motivation-Behavioral Skills Model: A general social psychological approach to understanding and promoting health behavior. In Suls, Wallston (Eds.), Social psychological foundations of health and illnes — https://www.wiley.com/en-us/Social+Psychological+Foundations+of+Health+and+Illness-p-9780631225157
- See also: Chang SJ, Choi S, Kim S, Song M. Intervention strategies based on Information-Motivation-Behavioral Skills Model for health behavior change: a systematic review. Asian Nurs Res 2014; 8: 172-81. — https://doi.org/10.1016/j.anr.2014.08.002
- See also: Kim YI, Park JS. Development and Evaluation of a Joint Health Self-management Program for the Elderly with Knee Osteoarthritis in Communities: Applying the IMB Model. J Korean Acad Community Health Nurs 2017; 28(1): 55-68. — https://synapse.koreamed.org/articles/1058496
- See also: To KW, Lee FKI. The effect of a theory-driven educational-intervention for improving adherence to inhalation therapy in patients with chronic obstructive pulmonary disease: A pilot study. Presented in Hong Kong College of Gerontology Nursing Scientifi — https://www.hkcgn.org/images/userfiles/newsletter/Newsletter_Issue28_8pp_r1.pdf
- See also: Matthews JNS. An introduction to randomized controlled clinical trials. London: Arnold, 2000. — https://books.google.com.hk/books/about/An_Introduction_to_Randomized_Controlled.html?id=0wrDQgAACAAJ&redir_esc=y
- See also: Kee JL. Laboratory and diagnostic tests with nursing implications, 6th ed.. Upper Saddle River, New Jersey: Prentice Hall, 2002. — https://www.amazon.com/Laboratory-Diagnostic-Tests-Nursing-Implications/dp/0130305197

DOCUMENTS (1):
  • Informed Consent Form (2021-08-04): https://cdn.clinicaltrials.gov/large-docs/11/NCT05008211/ICF_001.pdf